CLINICAL TRIAL: NCT03684993
Title: Effect of Gum Arabic (Acacia Gum) and Licorice (Glycyrrhiza Glabra) Mouthwashes Compared to Chlorhexidine Mouthwash on Caries Prevention and the Prevalence of Oral Side Effects in High Caries Risk Patients: A Randomized Controlled Clinical Trial
Brief Title: Caries Prevention and Side Effects of Gum Arabic and Licorice Extracts Versus Chlorhexidine in High Caries Risk Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Mohamed Kamal Eldin, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: arabic gum licorice CHX
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: High Caries Risk Patients; Caries; Antimicrobial Effect; Side Effect
MeSH Terms: interventions — Gum Arabic; Glycyrrhiza glabra extract; Chlorhexidine; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arabic gum extract (Experimental): natural product Arabic gum (acacia gum) prepared as a mouthwash
  Interventions: Drug: Arabic, Gum
- Licorice root extract (Experimental): natural product Licorice (Glycyrrhiza Glabra) root extract prepared as a mouthwash
  Interventions: Drug: Licorice Root
- Chlorhexidine (Active Comparator): chemical agent Chlorhexidine as a mouthwash
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Arabic, Gum — natural gum of acacia tree: Antimicrobial, anti-inflammatory medicinal plant used as a traditional oral hygiene substance (anticariogenic). It is used in treating sore throats, colds, bronchitis, toothache, gingival bleeding and mouth ulcers.
  Other Names: acacia gum
  Arms: Arabic gum extract
Drug: Licorice Root — natural licorice, herbal plant to relieve coughs, sore throats, and gastric inflammation. flavouring and sweetening agent. it's anti-caries, soothing anti-inflammatory and anticancer properties benefit against oral diseases and dental caries
  Other Names: Glycyrrhiza Glabra
  Arms: Licorice root extract
Drug: Chlorhexidine — chemical agent used as a mouthwash against cariogenic bacteria. considered the gold standard
  Other Names: Chlorhexidine gluconate or Chlorhexidine HCL
  Arms: Chlorhexidine

SUMMARY:
This trial is to test the caries prevention effect of Arabic gum and Licorice root extracts compared to Chlorhexidine in high caries risk patients. The antimicrobial efficacy and oral side effects from using these mouthwashes will also be tested.

DETAILED DESCRIPTION:
To evaluate the effect of Arabic gum (Acacia gum) and Licorice (Glycyrrhiza Glabra) mouthwashes in comparison to Chlorhexidine mouthwash on reducing caries incidence (development of new caries lesions), antimicrobial efficacy and the prevalence of oral side effects (adverse events) in high caries risk patients.

P: Population with high caries risk patients I1: Arabic Gum mouthwash I2: Licorice mouthwash C: Chlorhexidine mouthwash O1: (Primary outcome) incidence of new caries lesions O2: (secondary outcome) antimicrobial efficacy O3: oral side effects (adverse events) from mouthwash use

ELIGIBILITY:
Inclusion Criteria:

* High caries risk patients according to CAMBRA caries risk assessment tool
* Baseline of at least 2-3 active non-cavitated or cavitated carious lesionssz
* Baseline salivary Mutans streptococci count ≥ 106 CFU/ml
* Baseline salivary Lactobacilli count ≥ 104 CFU/ml
* Baseline DMF index of at least 3-5
* Cooperative patients approving to participate in the study

Exclusion Criteria:

* Any systemic conditions, severe medical complications
* Significant past or current medical condition that may affect oral health or oral flora
* Current medications (may affect the oral flora or salivary flow)
* Allergy to any of the ingredients of the study products
* Use of any antibiotics within the past 3 months
* Use of any mouth rinses within the past 3 months
* Current periodontitis (sites of probing pocket depth ≥ 5 mm)
* Evidence of parafunctional habits
* Dysfunction of temporomandibular joint
* Presence of developmental dental anomalies
* Presence of orthodontic appliance or removable prosthesis
* Pregnancy
* Xerostomia
* Heavy smoking
* Drug or alcohol addiction, or conditions that may decrease adhering to study protocol
* Lack of compliance

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Caries incidence - DMF index - visual and tactile clinical examination for caries detection according to the ICDAS critera | 1 year (detected after 3, 6, 9 and 12 months)
  development of new caries lesions. Clinical examination during study time to Measure DMF scoring index: any changes in number of decayed, missing and filled surfaces due to caries from baseline. Done according to International Caries Detection and Assessment System (ICDAS II criteria)

SECONDARY OUTCOMES:
Antimicrobial efficacy - Incubating agar plates - Colony forming units (CFU/mL) | 1 year (evaluated after 3, 6, 9 and 12 months)
  Antimicrobial effect against streptococcus mutans and lactocbacilli: saliva samples collected and total bacterial count measured after agar plates incubating, expressed in colony forming units
Side (Adverse) effect - subjective: Reporting Questionnaire - Binary outcome (yes/no) | 1 year (recorded after each month of mouthwash use)
  side effects from long term use of mouthwash

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta D, Gupta RK. Investigation of antibacterial efficacy of Acacia nilotica against salivary mutans streptococci: a randomized control trial. Gen Dent. 2015 Jan-Feb;63(1):23-7. PMID 25574715
- [Background] Hu CH, He J, Eckert R, Wu XY, Li LN, Tian Y, Lux R, Shuffer JA, Gelman F, Mentes J, Spackman S, Bauer J, Anderson MH, Shi WY. Development and evaluation of a safe and effective sugar-free herbal lollipop that kills cavity-causing bacteria. Int J Oral Sci. 2011 Jan;3(1):13-20. doi: 10.4248/IJOS11005. PMID 21449211
- [Background] Chandra Shekar BR, Nagarajappa R, Singh R, Thaku R. Antimicrobial efficacy of the combinations of Acacia nilotica, Murraya koenigii L. sprengel, Eucalyptus hybrid and Psidium guajava on primary plaque colonizers. J Basic Clin Pharm. 2014 Sep;5(4):115-9. doi: 10.4103/0976-0105.141954. PMID 25316992
- [Background] Almaz ME, Sonmez IS, Okte Z, Oba AA. Efficacy of a sugar-free herbal lollipop for reducing salivary Streptococcus mutans levels: a randomized controlled trial. Clin Oral Investig. 2017 Apr;21(3):839-845. doi: 10.1007/s00784-016-1827-y. Epub 2016 Apr 30. PMID 27129589
- [Background] Jain E, Pandey RK, Khanna R. Liquorice root extracts as potent cariostatic agents in pediatric practice. J Indian Soc Pedod Prev Dent. 2013 Jul-Sep;31(3):146-52. doi: 10.4103/0970-4388.117964. PMID 24021323